CLINICAL TRIAL: NCT03695029
Title: Maternal Screening and Antiviral Therapy in Pregnant Women to Reduce Mother-to-infant Transmission of Hepatitis B Virus
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 201010078M
Record Dates: First submitted 2018-09-20; First posted 2018-10-03 (Actual); Last update posted 2020-11-27 (Actual); Status verified 2020-11

CONDITIONS: Hepatitis B Virus Infection
MeSH Terms: conditions — Hepatitis B | interventions — tenofovir alafenamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- treatment group (Experimental): Pregnant women receiving tenofovir alafenamide 25 mg per day since 26-32 weeks of pregnancy to 2-4 weeks postpartum.
  Interventions: Drug: Tenofovir Alafenamide
- control group (No Intervention): control group receive no drug, only follow-up

INTERVENTIONS:
Drug: Tenofovir Alafenamide — Pregnant women receiving tenofovir alafenamide 25 mg per day since 26-32 weeks of pregnancy to 2-4 weeks postpartum.
  Arms: treatment group

SUMMARY:
To investigate the efficacy of using antiviral therapy in third trimester of pregnancy to reduce mother-to-infant HBV transmission, and to access the safety of such treatment for mothers and infants.

DETAILED DESCRIPTION:
This is a multi-centered study conducted in 12-16 collaborative hospitals in Taiwan, using tenofovir as antiviral therapy to reduce mother-to-infant transmission. The study group recruited pregnant women at 2nd to 3rd trimester receive tenofovir disoproxil fumurate (TDF) 2011-2018, June, and receive tenofovir alafenamide (TAF) 2018-2021. Control group did not receive antiviral treatment. Both group receive mother and infant follow-up up to 12 months after delivery.

ELIGIBILITY:
Inclusion criteria:

* Women aged 20-45 years in 28 to 32 weeks of pregnancy
* Positive HBsAg and HBeAg
* Serum viral load above 6 log10 IU/mL

Exclusion criteria:

* Major systemic disease of the mother or fetus
* Positive anti-HIV or anti-HCV
* Under treatment of antiviral therapy
* Pregnant woman whose ultrasonographic examination reveals congenital anomaly of the fetus
* Pregnant woman whose amniocentesis reveals any genetic abnormality

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Pregnant women
Enrollment: 120 (Estimated)
Dates: Start 2010-12-29 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Child HBsAg 6 mo | 6 months after delivery
  Serum status of HBsAg of the infants at 6 months old

SECONDARY OUTCOMES:
Child HBsAg 12 mo | 12 months after delivery
  Serum status of HBsAg of the infants at 12 months old
Maternal ALT elevation | 6 months after delivery
  Rate of postpartum maternal ALT elevation above 2X upper limit of normal within 6 months after delivery
Maternal HBeAg-seroconverion | 12 months after delivery
  HBeAg-seroconversion rate within 12 months after delivery
Maternal renal | 6 and 12 months post delivery
  Maternal serum creatinine (mg/dL) at 6 and 12 months post delivery
Materna bone marker | 6 and 12 months post delivery
  Maternal bone alkaline phosphatase (ug/L) at 6 and 12 months post delivery
Children's growth | 6 and 12 months after birth
  Children's growth: height (cm) in Z score at 6 and 12 months after birth
Children's growth | 6 and 12 months after birth
  Children's growth: weight (kg) in Z score at 6 and 12 months after birth

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

REFERENCES:
- [Derived] Chen HL, Lee CN, Chang CH, Lai MW, Tsai MC, Mu SC, Liu CJ, Shih JC, Wen WH, Hu RT, Huang CP, Hu KC, Chen CP, Lee CL, Chien RN, Chang KC, Hsu HY, Lee CC, Ni YH, Chang MH. Tenofovir alafenamide or tenofovir disoproxil fumarate in pregnancy to prevent HBV transmission: Maternal ALT trajectory and infant outcomes. Liver Int. 2024 Jun;44(6):1422-1434. doi: 10.1111/liv.15873. Epub 2024 Mar 8. PMID 38456620